CLINICAL TRIAL: NCT03986528
Title: Clinical Trial on the Survival Advantage of Kanglaite Injection (KLTi) in Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Clinical Trial of Kanglaite Injection (KLTi) in Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jie Li (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government); Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Jie Li, Chief of Medical Department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018YFC1707405
Record Dates: First submitted 2019-05-30; First posted 2019-06-14 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: NSCLC
Keywords: Advanced Non-Small Cell Lung Cancer; Kanglaite Injection; Chinese Herbal Medicine; Randomized Controlled Trial; Progression-free Survival
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kanglaite Injection + Chemotherapy (Experimental): Participants receive Kanglaite Injection PLUS first-line chemotherapy.
  Interventions: Drug: Kanglaite Injection+Chemotherapy
- Chemotherapy (Active Comparator): first-line chemotherapy.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Kanglaite Injection+Chemotherapy — Patients will receive investigator's choice of paclitaxel (135mg/m2 by IV infusion on Day 1 of each 21-28 day cycle) or pemetrexed (500mg/m2 by IV infusion on Day 1 of each 21-28 day cycle) or gemcitabine(1000mg/m2 by IV infusion on Days 1,8 of each 21-28 day cycle) PLUS cisplatin (75mg/m2 by IV infusion on Days 1 to 3 of each 21-28 day cycle) or carboplatin (AUC 6 by IV infusion on Days 1 of each 21-28 day cycle) according pathologic types. Patients with CR, PR, or SD after 4-6 cycles of platinum-based double chemotherapy regimens will receive non-platinum single-agent chemotherapy. The patients will also receive Kanglaite injection 200ml by IV infusion per day continuously for 14 days, commencing on the first day of chemotherapy.
  Arms: Kanglaite Injection + Chemotherapy
Drug: Chemotherapy — Patients will receive investigator's choice of paclitaxel (135mg/m2 by IV infusion on Day 1 of each 21-28 day cycle) or pemetrexed (500mg/m2 by IV infusion on Day 1 of each 21-28 day cycle) or gemcitabine(1000mg/m2 by IV infusion on Days 1,8 of each 21-28 day cycle) PLUS cisplatin (75mg/m2 by IV infusion on Days 1 to 3 of each 21-28 day cycle) or carboplatin (AUC 6 by IV infusion on Days 1 of each 21-28 day cycle) according pathologic types. Patients with CR, PR, or SD after 4-6 cycles of platinum-based double chemotherapy regimens will receive non-platinum single-agent chemotherapy.
  Arms: Chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Kanglaite Injection for advanced non-small cell lung cancer(NSCLC).

DETAILED DESCRIPTION:
This study include a multicenter, randomized, controlled post-market clinical trial.The randomized clinical trial will enroll approximately 334 patients. Participants will be randomly divided into experimental (n=167) and control groups (n=167).Patients in the experimental group will receive Kanglaite Injection combination with first-line chemotherapy based on NCCN Guidelines (2019.V3). Patients in the control group will receive first-line chemotherapy based on NCCN Guidelines (2019.V3).The primary endpoint is PFS(progression free survival).The research protocol was approved by the relevant ethics committees, and the study was conducted according to the Declaration of Helsinki and Good Clinical Practice guidelines. Patients gave written informed consent to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* A Histological or cytological confirmed diagnosis of Stage III-IV NSCLC, with no history of anticancer treatment including chemotherapy;
* Male or female aged 18-75years;
* Eastern Cooperative Oncology Group (ECOG) performance score 0-2;
* Life expectancy of at least 3 months;
* At least one radiographically measurable lesion per RECIST 1.1;
* Willing to join the clinic trail and sign informed consent;
* Able to comply with scheduled visits and treatments.

Exclusion Criteria:

* Presence of cerebral metastases;
* Confirmed positive for expression of expression of epidermal growth factor receptor (EGFR), activin receptor-like kinase (ALK), c-ros oncogene 1 (ROS1) mutation, or programmed death-ligand 1 (PD-L1)(tumor proportion score [TPS≥ 50%] in a genetic test;
* Participants with malignant pleural effusion underwent intrapleural injection chemotherapy;
* Current undergoing or preparing for treatment with target therapy;
* Current undergoing or preparing for radiotherapy to the thorax;
* Current undergoing or preparing treatment with tumor immunotherapy;
* Currently undergoing lipid-decreasing treament;
* Pregnant or breastfeeding woman;
* Fertile patients who are unwilling or unable to take effective contraceptive measures during the research period until 6 months after the study end later;
* A history of mental disorders；
* Severe and uncontrolled organic lesion or infection, including but not limited to cardiopulmonary failure and renal failure，which lead to poor tolerance of chemotherapy;
* Participated in other clinical trials of small molecule research drugs within 28 days prior to enrollment, or participated in other clinical trials of large molecule research drugs within 3 months before enrollment;
* Known allergy or intolerance to study medications;
* Considered to be otherwise unsuitable for the clinical study by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | Randomization until disease progression, death, or 12 months after randomized enrollment, whichever occurs first.
  Progression Free Survival (PFS), as Determined by the Investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Every two cycles (each cycle is 21-28 days) until disease progression, death, or 12 months after randomized enrollment, whichever occurs first.
  ORR is defined as the percentage of participants who had a Complete Response (CR:Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed by RECIST 1.1.
One-Year Survival Rate | Randomization until One year.
  One-year survival rate refers to the proportion of patients with a survival period of more than one year starting from randomized enrollment.
Quality of life of the patient | before and after each cycle of treatment, assessed up to 12 months after randomized enrollment
  This will be measured with validated questionnaires (EORTC-QLQ C30) and Lung Cancer Symptom Scale(LCSS).
Living ability of the patient | before and after each cycle of treatment, assessed up to 12 months after randomized enrollment
  This will be measured with validated questionnaires(ECOG) and Karnofsky performance status (KPS).
Blood lipid | every 41-56 days(2 cycles ) until disease progression, death, or assessed up to 12 months after randomized enrollment.
  total cholesterol, triacylglycerides, high density cholesterol, low density cholesterol.
Percentage of Participants With Adverse Events | Baseline until disease progression,death, or assessed up to 12 months after randomized enrollment.
  Percentage of Participants With Adverse Events in different arms.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Anhui Chest Hospital, Hefei, Anhui
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Gansu Provincial Tumor Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guanzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Academy of Traditional Chinese Medicine Affiliated Hospital, Changsha, Hunan
  - Hunan Provincial Tumor Hospital, Changsha, Hunan
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - XuZhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine,Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The Fourth Military Medical University Tangdu Hospital, Xian, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang Chinese Medicine University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
The results of the study will be issued to publications through scientific journals and conference reports. The anonymized datasets used and/or analyzed during the current study are available from the sponsor-investigator on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Gao R, Zhang Y, Hou W, Li J, Zhu G, Zhang X, Xu B, Wu Z, Wang H. Combination of first-line chemotherapy with Kanglaite injections versus first-line chemotherapy alone for advanced non-small-cell lung cancer: study protocol for an investigator-initiated, multicenter, open-label, randomized controlled trial. Trials. 2021 Mar 17;22(1):214. doi: 10.1186/s13063-021-05169-w. PMID 33731199